CLINICAL TRIAL: NCT02083952
Title: Impact of Swaddle Blanket on Gastroesophageal Reflux
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valley Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20131959
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Gastroesophageal Reflux; Apnea; Bradycardia; Oxygen Desaturations
MeSH Terms: conditions — Gastroesophageal Reflux; Apnea; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- swaddle blanket (Experimental)
  Interventions: Other: Swaddle Blanket

INTERVENTIONS:
Other: Swaddle Blanket — Two arms involve varying time spent in blanket

SUMMARY:
Gastroesophageal reflux disease (GERD) has been reported in up to 85% of all infants born prematurely, and has been associated with a wide range of symptoms. These include irritability, pauses in breathing, heart rate drops, declines in oxygen levels, chronic lung disease, and delays in growth and development. A novel approach to the mangement of GERD in infants is the use of an abdominal band, applying gentle pressure and possibly reducing the reflux of acid from the stomach. The purpose of this study is to evaluate the impact of a swaddle blanket with an abdominal band insert on the incidence of infant apnea, bradycardia, oxygen declines, and pH (acid) changes.

ELIGIBILITY:
Inclusion Criteria:

- NICU patients who have a 5 channel study requested by the attending neonatologist -

Exclusion Criteria:

-

Ages: 2 Days to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
pH | 24 hours
  all epochs of pH values below 4.0 will be measured

SECONDARY OUTCOMES:
apnea | 24 hours
  all breathing pauses greater than 20 seconds will be noted

OTHER OUTCOMES:
bradycardia | 24 hours
  all heart rate drops below 80 beats per minute will be noted
oxygen desaturations | 24 hours
  all oxygen drops below 92% will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Mary T Carbone, MD, Principal Investigator — The Valley Hospital
Locations (1):
- The Valley Hospital, Ridgewood, New Jersey, United States